CLINICAL TRIAL: NCT03843203
Title: Efficacy and Effectivity of Long Term Home Based tDCS in Fibromyalgia: an Explanatory Randomized Clinical Trial
Brief Title: Long Term Home Based tDCS in Fibromyalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Wolnei Caumo, Professor, M.D, PhD., Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-0330
Record Dates: First submitted 2018-01-17; First posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Fibromyalgia; Transcranial Direct Current Stimulation
Keywords: Pain; Brain derived neurotrophic factor; functional capacity
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Double-Blind, Randomized, Parallel Group, Sham-Controlled Clinical Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The researcher will receive equipment already programmed by a research assistant, so the researcher who will deliver the tDCS to perform stimulation will not know the programed stimulation. Patients will be instructed to discuss aspects of treatment with the respective investigator. Two independent evaluators who will not participate in the consultations where guidance on the use of tDCS will be provided will be trained to make outcome assessments in follow-up. Patients will not be aware of the type of intervention received, since the sham condition produces a stimulus, but no expected effects. In order to study the level of the blinding, at each moment of evaluation, the patient will be asked about the type of intervention that he / she believes to have received (active or simulated), and about the degree of safety in the response, using a standardized questionnaire. The blinding will be evaluated at the end of each treatment week by means of a standardized instrument.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- s-tDCS (Sham Comparator): - Intervention: 'Transcranial Direct Current Stimulation - tDCS The patients will receive tDCS sham treatment. The patients will receive sham tDCS treatment over primary motor cortex. According to 10-20 EEG system, anode will be placed at left C3 and cathode at o contralateral F3. In sham stimulation the device only release flow current, in the first 30 s of session and in the remaining 30s in the end of the session, during 20 minutes.
  Interventions: Device: Transcranial Direct Current Stimulation - tDCS
- M1 a-tDCS (Active Comparator): * Intervention: 'Transcranial Direct Current Stimulation - tDCS
  * The patients will receive tDCS active treatment over primary motor cortex.
  * According to 10-20 EEG system, anode will be placed at left C3 and cathode at contralateral supraorbital Fp2.
  * Active stimulation uses a 2 milliamperes current during 20 minutes.
  Interventions: Device: Transcranial Direct Current Stimulation - tDCS
- DLPFC a-tDCS (Active Comparator): * Intervention: 'Transcranial Direct Current Stimulation - tDCS
  * The patients will receive tDCS active treatment over dorsolateral prefrontal cortex.
  * According to 10-20 EEG system, anode will be placed at left F3 and cathode at contralateral F4.
  * Active stimulation uses a 2 milliamperes current during 20 minutes.
  Interventions: Device: Transcranial Direct Current Stimulation - tDCS

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation - tDCS — - Intervention: tDCS is a therapeutic method that modulates the membrane potential, where anodic stimuli induce cortical excitability and cathodic stimuli reduce it

SUMMARY:
Fibromyalgia(FM) is a widespread musculoskeletal pain syndrome characterized by fatigue, sleep disorders, cognitive impairment, depressive symptoms and neuro-vegetative symptoms. It is a multivariable and complex neurobiological process. FM worldwide prevalence according to American College of Rheumatology (ACR) 2010 diagnostic criteria is estimated under 5,4%. In USA the burden caused by FM is estimated at 29 billions every year, due to assistance, health care costs and retirement to loss of productivity. It is known that conventional pharmacological approaches present poor therapeutic response in more than 50% of these patients. It is conceivable that this limited results, at least in part, due to the lack of a complete elucidation of its pathophysiology.

Our hypothesis is that tDCS has a superior effect on clinical outcomes, functional capacity, cortical excitability, and psycho-affective functions compared to simulated treatment. In order to respond to the objectives of this study, a randomized, parallel-blinded clinical trial will be conducted. FM patients will be randomized to receive tDCS with anodic pole on the primary motor cortex and the cathode pole on the contralateral prefrontal cortex.

DETAILED DESCRIPTION:
Fibromyalgia(FM) is a widespread musculoskeletal pain syndrome characterized by fatigue, sleep disorders, cognitive impairment, depressive symptoms and neuro-vegetative symptoms. It is a multivariable and complex neurobiological process. FM worldwide prevalence according to ACR 2010 diagnostic criteria is estimated under 5,4%. In USA the burden caused by FM is estimated at 29 billions every year, due to assistance, health care costs and retirement to loss of productivity. It is known that conventional pharmacological approaches present poor therapeutic response in more than 50% of these patients. It is conceivable that this limited results, at least in part, due to the lack of a complete elucidation of its pathophysiology.

What is known so far is that the peripheral mechanisms contribute to the FM frame, but the central component surely commands the process, because the peripheral component does not explain ubiquitous fatigue, sleep problems, depressed mood and memory, catastrophic thinking, which are invariably as or more relevant than the pain of superficial structures. Diffuse hyperalgesia, allodynia, and the summation effect are added to the symptoms mentioned. Such symptoms are part of the central sensitization. Among dysfunctional FM processes, functional alterations of the motor cortex and its connections with subcortical structures that constitute the neuromatrix of pain have been demonstrated, as well as quantitative and qualitative alterations in fine sensitive fibers of the peripheral nervous system. Based on this complex nature of FM, the objective of this research is to obtain greater clarity about its pathophysiology and to identify distinctions between subgroups of patients with a view to advancing diagnosis and treatment, aiming at individualized therapy and improving outcomes, thereby attenuating , the significant loss to patients' lives and the heavy social and economic burden to patients and society.

As for the current therapeutic approach, in addition to drugs approved by the Food and Drug Administration (FDA) - duloxetine, milnacipran and pregabalin) the target has been techniques that may modify the dysfunctional neuroplasticity process, such as transcranial direct current stimulation tDCS) in order to counter-regulate the dysfunction responsible for triggering and maintaining FM symptoms. Although this technique is gaining space in the research and in the clinical scenario, many questions remain to be answered, such as: time of treatment, place to be stimulated (assembly method), how to perform maintenance therapy and benefit time after treatment, and, above all, which techniques could produce an additive effect (eg, physical activity, cognitive and pharmacological activity). From the presented scenario, the present project was organized, which is characterized as a clinical trial to evaluate the efficacy and the effectiveness of transcranial direct current stimulation (tDCS) and the dose (in the sessions) in the treatment of FM, with measures of pain, functional capacity and function of the descending pain modulator system as the outcomes. Also, potential predictors of (tDCS) response in primary outcomes will be: (a) Transcranial Magnetic Stimulation (TMS) parameters (motor evoked potential (MEP), intracortical inhibition (ICI), intracortical facilitation (ICF) and silent period (CSP)) ; (b) serum levels of brain-derived neurotrophic factor (BDNF) and its polymorphisms for the G (Val; / Met) alleles, as well as levels of the S100B protein; (c) level of central sensitization, catastrophism of pain and depressive symptoms.

In order to respond to the objectives of this study, a randomized, parallel-blinded clinical trial with 60 female patients with FM, diagnosed according to the criteria of the American Society of Rheumatology (2010 - revised in 2016), age between 19 and 65 years old, who will be randomized to receive tDCS with anodic pole on the primary motor cortex and the cathode pole on the contralateral prefrontal cortex. The sessions will last 20 min, the current intensity will be 2 milliamperes, with anodic pole on the primary motor cortex and the cathode pole on the dorsolateral prefrontal cortex of the left hemisphere. Patients will receive, in addition to training to administer home-based (tDCS) treatment, written instructions on physical exercises suggested by the investigator. The duration of treatment will be 8 weeks and a follow-up time after the end of the 12-week stimulation as recommended by the Initiative on Methods, Measurement and Pain Assessment in Clinical Trials (IMMPACT). Patients should respond daily to two questionnaires, one on the type of exercise performed and the duration of the exercises and another on the possible side effects of the tDCS. The home tDCS will be carried out with equipment developed by the research group coordinated by the proponent of this project, in partnership with the Biomedical Engineering of the Hospital of Clinics of Porto Alegre (HCPA), with a patent application with the National Institute of Industrial Property (INPI) under the number BR2020150164500. In addition to the possible contribution to knowledge production, this project aims to transfer the technology acquired and developed to the community, and in this way, it can benefit millions of people suffering from chronic FM pain with limited diagnostic and therapeutic perspective. In addition, to provide a cost-effective therapeutic technique for phase III studies on the use of large-scale home-based tDCS, a technique that can be extended to several neuropsychiatric conditions, such as depression and besides being able to assist as an adjuvant in the rehabilitation of sequelae of cerebral ischemia. Our hypothesis is that tDCS has a superior effect on clinical outcomes, functional capacity, cortical excitability, and psycho-affective functions compared to simulated treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women, who are able to read and write, with confirmed diagnosis of FM according to the criteria of the American College of Rheumatology (2010-2016).
* Pain score equal to or greater than six on the Numerical Pain Scale (NPS 0-10) on most days of the last 3 months.

Exclusion Criteria:

* Reside outside the Greater Porto Alegre area
* Pregnancy
* Contraindications to TMS and tDCS: metallic implant in the brain; medical devices implanted in the brain, cardiac pacemaker; cochlear implant;
* History of alcohol or drug abuse in the last 6 months; neurological diseases; history of head trauma or neurosurgery; decompensated systemic diseases, and chronic inflammatory diseases (lupus, rheumatoid arthritis, Sjogren's syndrome, Reiter's syndrome); uncompensated hypothyroidism; personal history of cancer, past or under treatment.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain level - first phase | 1 month
  Change from before and after the First phase of treatment on Pain scores assessed by a visual analogue scale (VAS 0 to 100mm) (0 means no pain - 100 means the worst pain imaginable)
Change in functional capacity - first phase | 1 month
  Change from before and after the First phase of treatment on Total score on the Brazilian Profile of Chronic Pain: Screen (BPCP:S) (range from 0 to 93; high numbers means more pain severity, interference in daily activities and emotional burden)

SECONDARY OUTCOMES:
Change in pain level - second phase | 3 months
  Change from before and after the Second phase of treatment on Pain scores assessed by a visual analogue scale (VAS 0 to 100mm) (0 means no pain - 100 means the worst pain imaginable)
Change in functional capacity - second phase | 3 months
  Change from before and after the First phase of treatment on Total score on the Brazilian Profile of Chronic Pain: Screen (BPCP:S) (range from 0 to 93; high numbers means more pain severity, interference in daily activities and emotional burden)
Change in Function of modulatory descending system | 1 month
  Change from before and after the First phase of treatment on the score in a numerical pain scale (NPS 0-10) for a moderate heat pain stimulus to the right arm (ventral region) during a conditioned pain modulation task (CPM-task), where participant keeps the counter-lateral hand in an iced cold water (0 to 1º Celsius)
Change in Function of corticospinal pathway | 1 month
  Change from before and after the First phase of treatment on measures of motor threshold (MT), motor evoked potential (MEP), intracortical facilitation (ICF), short intracortical inhibition (SICI), and cortical silent period (CSP) assessed with transcranial magnetic stimulation (TMS).
Change in levels of Brain derived neurotrophic factor - BDNF | 1 month
  Blood samples will be collected at baseline and after the First phase of intervention in order to determine BDNF serum levels using a standardized kit
Polymorphism of Brain derived neurotrophic factor - BDNF | 10 minutes
  Blood samples will be collected at baseline in order to determine BDNF gene polymorphism for the G allele (rs6265)

CONTACTS AND LOCATIONS:
Overall Officials: Wolnei Caumo, PhD, Study Director — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clauw DJ, Arnold LM, McCarberg BH; FibroCollaborative. The science of fibromyalgia. Mayo Clin Proc. 2011 Sep;86(9):907-11. doi: 10.4065/mcp.2011.0206. PMID 21878603
- [Background] Keeser D, Meindl T, Bor J, Palm U, Pogarell O, Mulert C, Brunelin J, Moller HJ, Reiser M, Padberg F. Prefrontal transcranial direct current stimulation changes connectivity of resting-state networks during fMRI. J Neurosci. 2011 Oct 26;31(43):15284-93. doi: 10.1523/JNEUROSCI.0542-11.2011. PMID 22031874
- [Background] Silva AF, Zortea M, Carvalho S, Leite J, Torres IL, Fregni F, Caumo W. Anodal transcranial direct current stimulation over the left dorsolateral prefrontal cortex modulates attention and pain in fibromyalgia: randomized clinical trial. Sci Rep. 2017 Mar 9;7(1):135. doi: 10.1038/s41598-017-00185-w. PMID 28273933
- [Background] Zanette SA, Dussan-Sarria JA, Souza A, Deitos A, Torres IL, Caumo W. Higher serum S100B and BDNF levels are correlated with a lower pressure-pain threshold in fibromyalgia. Mol Pain. 2014 Jul 8;10:46. doi: 10.1186/1744-8069-10-46. PMID 25005881
- [Derived] Lopes Alves R, Zortea M, Vicuna Serrano P, Laranjeira VDS, Franceschini Tocchetto B, Ramalho L, Fernanda da Silveira Alves C, Brugnera Tomedi R, Pereira de Almeida R, Machado Bruck S, Medeiros L, R S Sanches P, P Silva D Jr, Torres ILS, Fregni F, Caumo W. Modulation of neural networks and symptom correlated in fibromyalgia: A randomized double-blind multi-group explanatory clinical trial of home-based transcranial direct current stimulation. PLoS One. 2024 Nov 13;19(11):e0288830. doi: 10.1371/journal.pone.0288830. eCollection 2024. PMID 39536019
- [Derived] Caumo W, Lopes Ramos R, Vicuna Serrano P, da Silveira Alves CF, Medeiros L, Ramalho L, Tomeddi R, Bruck S, Boher L, Sanches PRS, Silva DP Jr, Ls Torres I, Fregni F. Efficacy of Home-Based Transcranial Direct Current Stimulation Over the Primary Motor Cortex and Dorsolateral Prefrontal Cortex in the Disability Due to Pain in Fibromyalgia: A Factorial Sham-Randomized Clinical Study. J Pain. 2024 Feb;25(2):376-392. doi: 10.1016/j.jpain.2023.09.001. Epub 2023 Sep 7. PMID 37689323
- [Derived] Serrano PV, Zortea M, Alves RL, Beltran G, Bavaresco C, Ramalho L, Alves CFDS, Medeiros L, Sanches PRS, Silva DP Jr, Lucena da Silva Torres I, Fregni F, Caumo W. The effect of home-based transcranial direct current stimulation in cognitive performance in fibromyalgia: A randomized, double-blind sham-controlled trial. Front Hum Neurosci. 2022 Nov 24;16:992742. doi: 10.3389/fnhum.2022.992742. eCollection 2022. PMID 36504629
- [Derived] Caumo W, Alves RL, Vicuna P, Alves CFDS, Ramalho L, Sanches PRS, Silva DP, da Silva Torres IL, Fregni F. Impact of Bifrontal Home-Based Transcranial Direct Current Stimulation in Pain Catastrophizing and Disability due to Pain in Fibromyalgia: A Randomized, Double-Blind Sham-Controlled Study. J Pain. 2022 Apr;23(4):641-656. doi: 10.1016/j.jpain.2021.11.002. Epub 2021 Nov 13. PMID 34785366